CLINICAL TRIAL: NCT02270567
Title: A Registry for Neuroendocrine Tumors
Brief Title: RegisterNET - A Registry for Neuroendocrine Tumors in the USA and Worldwide
Acronym: RegisterNET
Status: Enrolling by invitation | Type: Observational
Sponsor: Wren Laboratories LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: WREN_REGISTER_01
Record Dates: First submitted 2014-09-29; First posted 2014-10-21 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumor; Carcinoid; Neuroendocrine Carcinoma
Keywords: PRRT; Somatostatin Analogue; NETest; Progression; PPQ
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Carcinoma, Neuroendocrine; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood collection (RNA stabilization tube) used for neuroendocrine tumor biomarker measurements (NETest)
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: NETest — Non-invasive blood test
  Other Names: Multianalyte Algorithm Analysis of circulating neuroendocrine tumor transcripts

SUMMARY:
Neuroendocrine tumors are derived from the neuroendocrine system of the gastroenteropancreatic and bronchopulmonary tract systems. Treatment options include surgery, medical and ablative therapies as well as peptide-receptor radionuclide therapy. Survival is linked to early and accurate diagnoses or to the effective detection of disease recurrence and/or treatment failure. One challenge is to develop accurate non-invasive blood tests that can detect neuroendocrine tumor activity. A second challenge is to evaluate the effectiveness of molecular biomarkers in the natural history of this disease. RegisterNET registry aims at collecting data and blood samples from patients presenting with a NET. Data will be entered prospectively and anonymized after informed consent. All physicians who treat neuroendocrine tumor patients are invited to participate to the registry through prospective agreements and sub-study protocols with Wren Laboratories. Data will be evaluated within regular time frames, focusing on diagnostic accuracy for biomarkers in the different types and grades of tumors, treatment modalities and patient outcomes (e.g. disease recurrence and survival), thereby contributing to an understanding of the role of biomarkers in tumor management.

DETAILED DESCRIPTION:
Background: Survival for neuroendocrine tumors is linked to early and accurate diagnoses or to the effective detection of disease recurrence and/or treatment failure. Non-invasive biomarkers have been identified that can improve diagnosis and prognosis of patients. Little, however, is known about the utility of these markers in clinical practice.

Objective: To systematically and prospectively collect clinical information and blood samples for NETest from neuroendocrine tumors to evaluate the clinical validity of this biomarker for diagnosis, surveillance, and prediction of disease prognosis and response to targeted therapeutics.

Methods: All neuroendocrine tumors (gastroenteropancreatic and pulmonary) are following informed consent. Data will be entered prospectively and anonymized. Patient history including a quality of life survey are completed by contributing physicians and blood sample is collected for analysis. All information will be transferred to the database. Evaluation of treatment modalities and patient outcomes (e.g. disease recurrence) will be assessed at follow-up times.

The primary objectives of the project are to:

* monitor patients with neuroendocrine tumors
* provide descriptive statistical analyses
* assessment of diagnostic accuracy of NETest

The secondary objectives of the project include:

* assessment of disease recurrence, progression and prognosis
* analysis of patient survival

Analyses will include:

1. Descriptive statistical analyses including demographics, site, treatment, QoL assessment.
2. Clinical follow-up and blood chemistry results.
3. Correlation analyses between blood results e.g., changes in NETest and clinical data. This will include assessment of the time at which the blood chemistry results significantly (and consistently) increases and the time of tumor recurrence and an evaluation whether the change in blood results is predictive of disease recurrence or progression. Changes can also be used for prognosis and evaluating response to therapies e.g., PRRT.

ELIGIBILITY:
Inclusion Criteria:

* Gastroenteropancreatic neuroendocrine tumor
* Bronchopulmonary neuroendocrine tumor
* Gastroenteropancreatic neuroendocrine carcinoma
* Pre- and post-surgical patients
* Watch & Wait/no treatment
* Treatment including somatostatin analogues, PRRT, targeted therapies.
* Patient provides informed consent

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a histologically confirmed diagnosis of a neuroendocrine tumor undergoing treatment and follow-up evaluation. This includes real-world patients as well as patients included in investigator-initiated clinical studies (IICS) e.g., PRRT or curative surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-03 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Tumor-related recurrence or progression | 5 years
  Image-based identification of recurrent or progressive tumor disease
Tumor-related diagnosis | 1 year
  Histological confirmation of neuroendocrine tumor
Tumor-related mortality | 10 years
  Survival from disease

SECONDARY OUTCOMES:
Quality of Life Evaluation | 5 years
  Questionnaire to evaluate quality of life status
Biomarker prediction of treatment response and disease relapse | 10 years
  Biomarker prediction of treatment response and disease relapse. This involves measurements of changes in NETest levels between two time-points. Changes can be in actual values or be evaluated as % change. Alterations in blood measurements can be correlated with survival curves (PFS and/or OS).

CONTACTS AND LOCATIONS:
Locations (1):
- Wren Laboratories, Branford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identififed, anonymized information including changes in NETest and outcomes e.g., PFS.

REFERENCES:
- [Background] Modlin IM, Drozdov I, Kidd M. The identification of gut neuroendocrine tumor disease by multiple synchronous transcript analysis in blood. PLoS One. 2013 May 15;8(5):e63364. doi: 10.1371/journal.pone.0063364. Print 2013. PMID 23691035
- [Background] Modlin IM, Drozdov I, Kidd M. Gut neuroendocrine tumor blood qPCR fingerprint assay: characteristics and reproducibility. Clin Chem Lab Med. 2014 Mar;52(3):419-29. doi: 10.1515/cclm-2013-0496. PMID 24127543
- [Background] Modlin IM, Drozdov I, Alaimo D, Callahan S, Teixiera N, Bodei L, Kidd M. A multianalyte PCR blood test outperforms single analyte ELISAs (chromogranin A, pancreastatin, neurokinin A) for neuroendocrine tumor detection. Endocr Relat Cancer. 2014 Aug;21(4):615-28. doi: 10.1530/ERC-14-0190. PMID 25015994
- [Background] Modlin IM, Drozdov I, Bodei L, Kidd M. Blood transcript analysis and metastatic recurrent small bowel carcinoid management. BMC Cancer. 2014 Aug 5;14:564. doi: 10.1186/1471-2407-14-564. PMID 25095873
- [Result] Kidd M, Drozdov IA, Chirindel A, Nicolas G, Imagawa D, Gulati A, Tsuchikawa T, Prasad V, Halim AB, Strosberg J. NETest(R) 2.0-A decade of innovation in neuroendocrine tumor diagnostics. J Neuroendocrinol. 2025 Apr;37(4):e70002. doi: 10.1111/jne.70002. Epub 2025 Feb 13. PMID 39945192
- [Result] Liu E, Paulson S, Gulati A, Freudman J, Grosh W, Kafer S, Wickremesinghe PC, Salem RR, Bodei L. Assessment of NETest Clinical Utility in a U.S. Registry-Based Study. Oncologist. 2019 Jun;24(6):783-790. doi: 10.1634/theoncologist.2017-0623. Epub 2018 Aug 29. PMID 30158287
- [Derived] Kidd M, Kitz A, Drozdov I, Modlin I. Neuroendocrine Tumor Omic Gene Cluster Analysis Amplifies the Prognostic Accuracy of the NETest. Neuroendocrinology. 2021;111(5):490-504. doi: 10.1159/000508573. Epub 2020 May 11. PMID 32392558